CLINICAL TRIAL: NCT05339555
Title: IUD Self-Removal: A Study to Pilot the Feasibility of a Novel Technique
Brief Title: IUD Self-Removal Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Jessica Reid, Clinical Instructor, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00023967
Record Dates: First submitted 2022-04-15; First posted 2022-04-21 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: IUD
Keywords: IUD Removal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- IUD Self-Removal (Other)
  Interventions: Other: Instructions for IUD Self-Removal Provided to Participant

INTERVENTIONS:
Other: Instructions for IUD Self-Removal Provided to Participant — The provider will offer any individual presenting for in-person IUD removal or exchange (removal-replacement) the option for self-removal. The participant will be provided a 'how to' instruction sheet with information on positioning and what to expect. The participant will first attempt removal with clean hands if desired, then utilizing non-sterile, clean gloves (not explicitly tested in prior studies) and if that fails, the use of a menstrual cup (a novel technique). If not successful, the provider will perform standard IUD removal in the clinic.

SUMMARY:
This is a pilot study designed to test the effectiveness of several techniques for intrauterine device (IUD) self-removal and to understand patient preferences regarding IUD self-removal and indicators of success as well as understanding the impacts of IUD self-removal on other clinical care.

DETAILED DESCRIPTION:
The Investigators propose to test a novel method for self-removal of IUDs in an effort to increase the proportion of patients who are able to successfully and safely remove their IUD when desired. Participants will attempt self-removal in office, where a provider will be able to remove the IUD if unsuccessful. Participants will be instructed on current and novel techniques and the investigators will examine indicators of success as well as patient and provider preferences.

ELIGIBILITY:
Inclusion Criteria:

* Presenting at clinic for IUD removal or exchange
* Willing and able to give consent with literacy in English or Spanish

Exclusion Criteria:

* Participants who are referred for a complicated IUD removal such as a stingless IUD, prior failed IUD removal attempt, or an IUD failure.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-06-10 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of IUD Self-Removal Techniques | Immediately after IUD Removal
  Proportion of participants who successfully remove their IUDs

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Reid, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science Univeristy, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No